CLINICAL TRIAL: NCT03179033
Title: Impact of Fluid and Passive Leg Raising on Cardiac Output in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-16-3259-ER-CTIL
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-06

CONDITIONS: Artificial Heart Device User
Keywords: LVAD; Passive leg raising

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Left Ventricular Assist Device (LVAD) implantation is a common surgical procedure in patients with end-stage heart failure. Optimal fluid management is essential for adequate postoperative treatment. It is important to identify which patients will benefit from fluid administration. Passive leg raising (PLR) is a validated dynamic method to predict fluid responsiveness in patients with heart failure by inducing a transient increase in cardiac preload. Objective: To investigate the role of PLR on the management of patients following LVAD implantation in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients after VAD implantation

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure candidate for assist device implantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Responsiveness to passive leg raising in patients early after LVAD implantation | 5 minutes
  Change in LVAD flow due to passive leg raising

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel